CLINICAL TRIAL: NCT03011801
Title: Reducing Fetal Exposure to Maternal Depression to Improve Infant Risk Mechanisms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); University of Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MH109662; R01MH109662 (NIH)
Record Dates: First submitted 2017-01-04; First posted 2017-01-05 (Estimated); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Behavioral: Interpersonal Therapy (Experimental): Individual psychotherapy that includes an initial engagement session and a total of 8 sessions. IPT focuses on psychoeducation and interpersonal skill building to decrease interpersonal conflict and increase interpersonal support and competence.
  Interventions: Behavioral: Interpersonal Therapy
- Enhanced Usual Care (Placebo Comparator): Maternity support services (MSS) is the usual standard of care for pregnant women. A multi-disciplinary team of obstetric care providers routinely screen women for possible depression diagnosis. If a woman screens positive, she is seen by a behavioral health specialist (BHS) for further assessment and to initiate treatment, if necessary. The goals of MSS include offering services to promote healthy pregnancies and positive birth and parenting outcomes, including integrating mental health and prenatal care. Women with elevated depressive symptoms are seen by BHS throughout the pregnancy and postpartum period and then bridged to mental health treatment. BHS provides eclectic-based care but does not provide IPT.
  Interventions: Behavioral: Enhanced usual care

INTERVENTIONS:
Behavioral: Interpersonal Therapy — reducing conflict in relationships, increasing social support in relationships, improving communication, reducing depressive symptoms
  Other Names: IPT
  Arms: Behavioral: Interpersonal Therapy
Behavioral: Enhanced usual care — Treatment as Usual, including eclectic and supportive therapy, as well as psychiatric medication
  Other Names: Maternity Support Services (MSS)
  Arms: Enhanced Usual Care

SUMMARY:
This study evaluates Interpersonal Therapy (IPT) in the treatment of depression among pregnant women with elevated depressive symptoms. Half of the women will be randomized to receive IPT, and the other half will get Treat As Usual, provided via behavioral health in the hospital.

DETAILED DESCRIPTION:
Exposure to maternal depressive symptoms is one of the most well established risk factors for the development of later child psychopathology. Accumulating evidence from naturalistic observational studies documents that fetal exposure to maternal depressive symptoms is associated with risk for later child mental health problems. Maternal depression is one of the most common prenatal complications with approximately 40% of women experiencing elevated levels of depressive symptoms. The majority of past research has been correlational, so potential causal conclusions have been limited. This project will break new ground by testing the hypothesis that manipulating maternal depressive symptoms will benefit infant outcomes. In this project, maternal depressive symptoms will be reduced using brief interpersonal therapy (IPT), a well-established and efficacious treatment, and testing whether this reduction leads to an improvement in the development of infant mechanisms associated with risk for later psychopathology. The investigators propose to assess 300 pregnant women who report elevated levels of depressive symptoms and their infants. Prior to the intervention, maternal measures of depressive symptoms will be collected. Then half of the women will be randomized to receive IPT and the other half will receive enhanced usual care (TAU). After completion of the intervention, maternal measures will be collected longitudinally through 14 months postpartum. Infants will be evaluated at birth and two other times. Infants will be assessed across four units of analysis (brain structure and function, physiology, behavior, and maternal-report).

ELIGIBILITY:
Inclusion Criteria:

* Adult women (over 18 years of age)
* A singleton intrauterine pregnancy
* English speaking
* Elevated depressive symptoms based on screening with the Edinburgh Postnatal Depression Scale (EPDS) with score > 9

Exclusion Criteria:

* Bipolar disorder and psychosis based on the Structured Clinical Interview for DSM-IV Axis I Disorders (SCID-NP)
* Current psychotropic medication use or current CBT/IPT usage
* An HPA axis or an endocrine disorder
* Maternal substance use [assessed using maternal report and urine toxicology
* Corticosteroid medication use during this pregnancy
* Invitto fertilization
* Presence of cervical or uterine abnormalities

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2024-05-28 (Actual)

PRIMARY OUTCOMES:
Presence of a Major Depressive Episode on SCID interview | 12 months post pregnancy
  Presence of a depression diagnosis as measured by a semi-structured diagnostic evaluation
Symptom Checklist 20 (SCL20) | post intervention (approximately 2-3 months post baseline)
  Self reported Depression Scores. higher scores=more depression
Symptom Checklist 20 (SCL20) | 6 months post intervention
  Self reported Depression Scores. higher scores=more depression
Symptom Checklist 20 (SCL20) | 12 months post intervention
  Self reported Depression Scores. higher scores=more depression

SECONDARY OUTCOMES:
Edinburgh Postnatal Depression Scale (EPDS) | post intervention (approximately 2-3 months post baseline)
  Self reported Depression Scores. higher scores=more depression
Edinburgh Postnatal Depression Scale (EPDS) | 6 months post intervention
  Self reported Depression Scores. higher scores=more depression
Edinburgh Postnatal Depression Scale (EPDS) | 12 months post intervention
  Self reported Depression Scores. higher scores=more depression
Work and Social Adjustment Scale (WSAS) | post intervention (approximately 2-3 months post baseline)
  general maternal functioning
Work and Social Adjustment Scale (WSAS) | 6 month post intervention
  general maternal functioning
Work and Social Adjustment Scale (WSAS) | 12 month post intervention
  general maternal functioning

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin L Hankin, PhD, Principal Investigator — University of Illinois Urbana Champaign; Elysia P Davis, PhD, Principal Investigator — University of Denver
Locations (2):
- United States (2):
  - University of Denver, Denver, Colorado
  - University of Illinois, Urbana, Illinois

IPD SHARING:
Plan to Share IPD: Yes
NIMH Data Archive
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: 1 year after publication of relevant paper in refereed journal
Access Criteria: appropriate, reasonable scientific request to co-PIs

REFERENCES:
- [Derived] Davis EP, Demers CH, Deer L, Gallop RJ, Hoffman MC, Grote N, Hankin BL. Impact of prenatal maternal depression on gestational length: post hoc analysis of a randomized clinical trial. EClinicalMedicine. 2024 Apr 22;72:102601. doi: 10.1016/j.eclinm.2024.102601. eCollection 2024 Jun. PMID 38680516
- [Derived] Hankin BL, Demers CH, Hennessey EP, Perzow SED, Curran MC, Gallop RJ, Hoffman MC, Davis EP. Effect of Brief Interpersonal Therapy on Depression During Pregnancy: A Randomized Clinical Trial. JAMA Psychiatry. 2023 Jun 1;80(6):539-547. doi: 10.1001/jamapsychiatry.2023.0702. PMID 37074698